CLINICAL TRIAL: NCT00407602
Title: Argus® II Retinal Stimulation System Feasibility Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Sight Medical Products (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-003-001; National Eye Institute (NEI) (Other Grant/Funding Number: 2R01EY012893-06A1)
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2021-12-30 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; device; retinal implant; retinal prosthesis; RP; outer retinal degeneration
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implant of Argus II Retinal Prosthesis (Other): This is a single group study where the status and performance of the implanted eye prior to surgery serves as the comparator.
  Interventions: Device: Implant of Argus II Retinal Prosthesis

INTERVENTIONS:
Device: Implant of Argus II Retinal Prosthesis — epiretinal implantation of device

SUMMARY:
Investigational Phase of the Study:

The objective of this feasibility study is to evaluate the safety and utility of the Argus II Retinal Stimulation System in providing visual function to blind subjects with retinitis pigmentosa.

Post-Approval Phase of the Study:

To collect post-approval data in order to monitor the ongoing safety and reliability of the Argus II System

DETAILED DESCRIPTION:
During the post-approval phase, subjects will undergo annual eye exams, assessments of medical status and adverse events, and measurement of stimulation thresholds. In addition, at the mutual agreement of the investigator and the subject, subjects will have the option of participating in psychophysical research which could occur as frequently as monthly. Functional tests at 10 years: photographic flash, square localization, direction of motion and grating visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed history of retinitis pigmentosa (all centers) or outer retinal degeneration (France, U.K., Switzerland, Mexico only) with remaining visual acuity of bare light perception (all centers) or 2.3 logMAR (France, U.K., Switzerland, Mexico only) or worse in both eyes.
* Functional ganglion cells and optic nerve as determined by a measurable electrically evoked response or documented light perception.
* A history of former useful form vision in the worse-seeing eye.
* Must be at least the following age at the time of enrollment: 25 (USA, Switzerland) or 18 (France, U.K., and Mexico) years old
* Must reside within 2 hours (USA, UK and Mexico) or 3 hours (France and Switzerland) distance (by ground transportation) of the investigational site.
* Must be willing and able to comply with the protocol testing and follow-up requirements.

Exclusion Criteria:

* Optic Nerve disease

  * History of glaucoma
  * Optic neuropathy or other confirmed damage to optic nerve or visual cortex damage
* Diseases or conditions that effect retinal function including but not limited to:

  * Central retinal artery/vein occlusion (CRAO or CRVO)
  * End-stage diabetic retinopathy
  * Retinal detachment or history of retinal detachment
  * Trauma
  * Infectious or inflammatory retinal diseases
* Diseases or conditions that prevent adequate visualization of the retina including, but not limited to corneal degeneration that cannot be resolved before implant.
* Diseases or conditions of the anterior segment that prevent the ability to adequately perform the physical examination including but not limited to trauma or lid malpositions.
* Diseases of the ocular surface including but not limited to keratitis sicca.
* An ocular condition that predisposes the subject to eye rubbing.
* Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

  * Cognitive decline including diagnosed forms of dementia and/or progressive neurological disease
  * Psychiatric Disease including diagnosed forms of depression
  * Does not speak a principal language associated with the region
  * Deafness or selective frequency hearing loss that prevents hearing device alarms and alerts.
* Pregnancy
* Subject has another active implantable device (e.g. cochlear implant), or any form of metallic implant in the head
* Conjunctival thinning which may predispose the subject to conjunctival erosion in the area where the implant will be installed extra-ocularly.
* Subject is participating in another investigational drug or device study that may conflict with the objectives, follow-up or testing of this study
* Any health concern that makes general anesthesia inadvisable.
* Subject has unrealistic expectations of the implant.
* Known allergy or contraindication to anticipated pre-operative, intra-operative or post-operative medications.
* Conditions likely to limit life to less than 1 year from the time of screening.
* Diseases or conditions that, in the judgement of the surgeon, impede the ability to implant the device or would prevent the system from functioning for the duration of the study (e.g. strabismus)
* Axial eye length <21.5 mm or >26.0 mm in the implanted eye as measured by ultrasound (US only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Ripley, Study Director — Second Sight Medical Products
Locations (12):
- United States (7):
  - Doheny Eye Institute, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins, Wilmer Eye Institute, Baltimore, Maryland
  - Columbia University, Department of Ophthalmology, Edward S. Harkness Eye Institute, New York, New York
  - University of Pennsylvania, Scheie Eye Institute, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas
- Centre d'Investigation Clinique, Service d'Ophtalmologie, Quinze-Vingts National Eye Hospital, 28 rue de Charenton, 75557 Cedex 12, Paris, France
- Puerta de Hierro, Centro Medico, Centro de Retina, Zapopan, Jalisco, Mexico
- Clinique d'Ophthalmologie Hopitaux, Universitaires de Geneve 22 rue Alcide Jentzer 1205, Geneva, Switzerland
- United Kingdom (2):
  - Moorfields Eye Hospital, Vitreoretinal Research Unit, London
  - Manchester Royal Eye Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiland JD, Faraji B, Greenberg RJ, Humayun MS, Shellock FG. Assessment of MRI issues for the Argus II retinal prosthesis. Magn Reson Imaging. 2012 Apr;30(3):382-9. doi: 10.1016/j.mri.2011.12.005. Epub 2012 Jan 20. PMID 22260934
- [Result] Humayun MS, Dorn JD, da Cruz L, Dagnelie G, Sahel JA, Stanga PE, Cideciyan AV, Duncan JL, Eliott D, Filley E, Ho AC, Santos A, Safran AB, Arditi A, Del Priore LV, Greenberg RJ; Argus II Study Group. Interim results from the international trial of Second Sight's visual prosthesis. Ophthalmology. 2012 Apr;119(4):779-88. doi: 10.1016/j.ophtha.2011.09.028. Epub 2012 Jan 11. PMID 22244176
- [Result] Barry MP, Dagnelie G; Argus II Study Group. Use of the Argus II retinal prosthesis to improve visual guidance of fine hand movements. Invest Ophthalmol Vis Sci. 2012 Aug 1;53(9):5095-101. doi: 10.1167/iovs.12-9536. PMID 22661464
- [Result] Ahuja AK, Dorn JD, Caspi A, McMahon MJ, Dagnelie G, Dacruz L, Stanga P, Humayun MS, Greenberg RJ; Argus II Study Group. Blind subjects implanted with the Argus II retinal prosthesis are able to improve performance in a spatial-motor task. Br J Ophthalmol. 2011 Apr;95(4):539-43. doi: 10.1136/bjo.2010.179622. Epub 2010 Sep 29. PMID 20881025
- [Derived] Arevalo JF, Al Rashaed S, Alhamad TA, Al Kahtani E, Al-Dhibi HA; KKESH Collaborative Retina Study Group. Argus II retinal prosthesis for retinitis pigmentosa in the Middle East: The 2015 Pan-American Association of Ophthalmology Gradle Lecture. Int J Retina Vitreous. 2021 Oct 27;7(1):65. doi: 10.1186/s40942-021-00324-6. PMID 34706764
- [Derived] Sabbah N, Authie CN, Sanda N, Mohand-Said S, Sahel JA, Safran AB. Importance of eye position on spatial localization in blind subjects wearing an Argus II retinal prosthesis. Invest Ophthalmol Vis Sci. 2014 Nov 20;55(12):8259-66. doi: 10.1167/iovs.14-15392. PMID 25414187
- [Derived] Ahuja AK, Yeoh J, Dorn JD, Caspi A, Wuyyuru V, McMahon MJ, Humayun MS, Greenberg RJ, Dacruz L. Factors Affecting Perceptual Threshold in Argus II Retinal Prosthesis Subjects. Transl Vis Sci Technol. 2013 Apr;2(4):1. doi: 10.1167/tvst.2.4.1. Epub 2013 Apr 12. PMID 24049718
- [Derived] de Juan E Jr, Spencer R, Barale PO, da Cruz L, Neysmith J. Extraction of retinal tacks from subjects implanted with an epiretinal visual prosthesis. Graefes Arch Clin Exp Ophthalmol. 2013 Oct;251(10):2471-6. doi: 10.1007/s00417-013-2452-y. Epub 2013 Sep 8. PMID 24013578
- [Derived] Stronks HC, Barry MP, Dagnelie G. Electrically elicited visual evoked potentials in Argus II retinal implant wearers. Invest Ophthalmol Vis Sci. 2013 Jun 6;54(6):3891-901. doi: 10.1167/iovs.13-11594. PMID 23611993
- [Derived] Dorn JD, Ahuja AK, Caspi A, da Cruz L, Dagnelie G, Sahel JA, Greenberg RJ, McMahon MJ; gus II Study Group. The Detection of Motion by Blind Subjects With the Epiretinal 60-Electrode (Argus II) Retinal Prosthesis. JAMA Ophthalmol. 2013 Feb;131(2):183-9. doi: 10.1001/2013.jamaophthalmol.221. PMID 23544203
- [Derived] Ahuja AK, Behrend MR. The Argus II retinal prosthesis: factors affecting patient selection for implantation. Prog Retin Eye Res. 2013 Sep;36:1-23. doi: 10.1016/j.preteyeres.2013.01.002. Epub 2013 Mar 14. PMID 23500412
- [Derived] Olson JL, Velez-Montoya R, Mandava N, Stoldt CR. Intravitreal silicon-based quantum dots as neuroprotective factors in a model of retinal photoreceptor degeneration. Invest Ophthalmol Vis Sci. 2012 Aug 17;53(9):5713-21. doi: 10.1167/iovs.12-9745. PMID 22761263
- [Derived] Perez Fornos A, Sommerhalder J, da Cruz L, Sahel JA, Mohand-Said S, Hafezi F, Pelizzone M. Temporal properties of visual perception on electrical stimulation of the retina. Invest Ophthalmol Vis Sci. 2012 May 4;53(6):2720-31. doi: 10.1167/iovs.11-9344. PMID 22447863

RESULTS

PARTICIPANT FLOW:
Groups:
- Implant of Argus II Retinal Prosthesis: This is a single group study where the status and performance of the implanted eye prior to surgery serves as the comparator.
  Argus II Retinal Stimulation System: epiretinal implantation of device
Period: Overall Study
Arm/Group | Implant of Argus II Retinal Prosthesis
Started | 30
Completed | 23
Not Completed | 7
Not completed — Death - unrelated to device | 1
Not completed — Device explanted | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Implant of Argus II Retinal Prosthesis
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 58.3 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14
  United Kingdom | 10
  France | 4
  Switzerland | 2

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Grating Visual Acuity is performed at Baseline and at various timepoints throughout the study. As of the 10 year final testing, the total number of subjects that were able to score on the logMAR scale are indicated below. The device has a scale from 1.6 to 2.9 logMAR. Maximum likelihood estimation of visual acuity is based on BEST-PEST algorithm.
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm: Only one arm in this study, treatment arm.
Arm/Group | Single Arm
Number analyzed (Participants) | 13
Participants | 2

2. Primary Outcome: Number of Participants With Adverse Events
Description: Evaluate ocular adverse events reported for all subjects from day of implant through 10 years of study participation
Time Frame: 10 years
Measure: Number; unit: participants
Groups:
- Single Arm: Single arm with fellow eye as comparator
Arm/Group | Single Arm
Number analyzed (Participants) | 30
participants
  Total number of subjects with serious ocular AEs | 13
  Total number of subjects with non-serious ocular AEs | 28

3. Secondary Outcome: Massof Activity Inventory
Description: The Massof Activity Inventory measures changes in ability to perform activities of daily living in terms of Goals and Tasks in logits (log-odds units). A logit scale is an equal interval linear scale that represents probability values in terms of real numbers. There is no minimum or maximum scale used in this testing. In this case, a Rasch distribution (using an Andrich rating model) was used to find the maximum likelihood of difficulty of achieving Goals and Tasks, represented in logits. The change in mean logit value between baseline and the 36Month visit for each subject are provided below along with the 95% confidence interval (CI) for the change. A positive change in the Goals or Tasks score which is greater than 0.2 (with a CI less than the mean logit value), is interpreted as a clinically significant increase in functional ability (better outcome).
Time Frame: 3 years
Population: Data for all 14 US subjects analyzed
Measure: Mean (95% Confidence Interval); unit: Logit scale
Arm/Group | Implant of Argus II Retinal Prosthesis
Number analyzed (Participants) | 14
Logit scale
  Subject1-Goals | -0.1 [-.87 to 0.67]
  S2-Goals | 1.0 [0.18 to 1.82]
  S3-Goals | 0.3 [-0.33 to 0.93]
  S4-Goals | 0.1 [-0.67 to 0.87]
  S5-Goals | 0.1 [-0.76 to 0.96]
  S6-Goals | -0.2 [-0.8 to 0.4]
  S7-Goals | -1.6 [-2.32 to -0.88]
  S8-Goals | 0.9 [0.21 to 1.59]
  S9-Goals | 0.2 [-0.25 to 0.65]
  S10-Goals | -0.3 [-0.86 to 0.26]
  S11-Goals | 0.1 [-0.51 to 0.71]
  S12-Goals | 0.0 [-0.57 to 0.57]
  S13-Goals | 0.5 [-0.16 to 1.16]
  S14 -Goals | NA [NA to NA] — Error in test administration, data determined to be invalid.
  S1-Tasks | 0.4 [-0.19 to 0.99]
  S2-Tasks | -0.2 [-0.45 to 0.05]
  S3-Tasks | 0.4 [0.16 to 0.64]
  S4-Tasks | -0.1 [-0.46 to 0.26]
  S5-Tasks | 0.6 [0.14 to 1.06]
  S6-Tasks | 0.2 [-0.06 to 0.46]
  S7-Tasks | -0.3 [-0.81 to 0.21]
  S8-Tasks | 2.0 [1.52 to 2.48]
  S9-Tasks | 0.8 [-0.09 to 1.69]
  S10-Tasks | -0.4 [-0.71 to -0.09]
  S11-Tasks | -0.2 [-0.45 to 0.05]
  S12-Tasks | -0.3 [-0.62 to 0.02]
  S13-Tasks | 0.2 [-0.11 to 0.51]
  S14-Tasks | NA [NA to NA] — Error in test administration, data determined to be invalid.

4. Secondary Outcome: Quality of Life - Tasks for Daily Living
Description: Quality of life is being measured using the VisQOL survey. This instrument, developed by researchers at the University of Melbourne, Australia, is a vision and quality of life-related utility measure intended to evaluate healthcare interventions for the visually impaired. The utility score is a preference-based measure of vision-related quality of life (Dimension 7 score (Health Dimension Score (1=Best, 0=Worst)). It measures subjective quality of life on a scale of 0 to 1, where 0 represents worst possible quality of life and 1 represents perfect quality of life.
Time Frame: 3 years
Population: 30 subjects were analyzed comparing Baseline visit to the last visit when VisQOL was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Implant of Argus II Retinal Prosthesis
Number analyzed (Participants) | 30
units on a scale | .6191 (.2146)

5. Secondary Outcome: Orientation and Mobility
Description: Argus II System for orientation and mobility, each subject completed two tests (walking to a high-contrast "door" on the wall and following a straight line on the floor) at various timepoints throughout the study. Accuracy (percent of trials where the subject successfully reached the target) was measured with the device system ON and system OFF. Average % success rates across the analysis population are provided for each modality and for each test at the 60 month time point.
Time Frame: 5 years
Population: Data for all 14 US subjects analyzed
Measure: Mean (Standard Deviation); unit: percentage of successful trials
Arm/Group | Single Arm
Number analyzed (Participants) | 14
percentage of successful trials
  Average % system ON-Door Task | 58 (24)
  Average % system OFF-Door Task | 18 (19)
  Average % system ON-Line Task: number analyzed (Participants) | 13
  Average % system ON-Line Task | 68 (36)
  Average % system OFF-Line Task: number analyzed (Participants) | 13
  Average % system OFF-Line Task | 10 (13)

6. Secondary Outcome: Visual Function
Description: Square localization (SL) and Direction of Motion (DOM) testing performed at specific protocol intervals. SL tests ability of subjects to locate high-contrast square on black screen. DOM tests ability of subjects to determine the direction a white bar is moving over a black screen. Each test is performed with the system ON and then compared to performance with the system OFF. Number of subjects who performed significantly better with the system ON is indicated below.
Time Frame: 10 years
Population: Data available only on 13 of the 14 US subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Implant of Argus II Retinal Prosthesis
Number analyzed (Participants) | 13
Participants
  SL - Number of subjects with significantly better with system ON | 9
  DOM - Number of subjects with significantly better with system ON | 4

7. Secondary Outcome: Stability of Implant - 5 Years Post Implant
Description: Stability of electrode array on the retina. Qualitative review of imaging: retinal and array landmarks compared from all time points post implant.
Time Frame: 5 years
Population: Data for all 14 US subjects analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Implant of Argus II Retinal Prosthesis
Number analyzed (Participants) | 14
Participants
  Stable position of array on Array position stable-no rotation | 8
  Minor array rotation | 5
  Inconclusive data | 1

8. Secondary Outcome: Device Reliability
Description: Number of participants with functional devices 10 years post implant
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Implant of Argus II Retinal Prosthesis
Number analyzed (Participants) | 30
Participants | 28

ADVERSE EVENTS:
Time Frame: 10 years
Description: Ocular events are reportable for this protocol from day of implant through the last study visit for each subject.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=30)
Conjunctival dehiscence (Eye disorders) | 4 (4)
Conjunctival erosion (Eye disorders) | 6 (9)
Corneal melt (Eye disorders) | 1 (1)
Endophthalmitis - infective (Eye disorders) | 4 (4)
Epiretinal membrane (Eye disorders) | 1 (1)
Hypotony (Eye disorders) | 5 (5)
Iris rubeosis (Eye disorders) | 1 (1)
Keratitis - infective (Eye disorders) | 1 (1)
Migration (extra-ocular) of intraocular silicone oil (Eye disorders) | 1 (1)
Re-tack (Eye disorders) | 2 (2) — Re-tack to hold the device in place on the retina
Retinal detachment - rhegmatogenous (Eye disorders) | 3 (3)
Retinal detachment - tractional and serous (Eye disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=30)
360 Circumferential Vitreous Band Traction (Eye disorders) | 1 (1)
Choroidal detachment (Eye disorders) | 6 (6)
Choroidal effusion (Eye disorders) | 1 (1)
Conjunctival congestion (Eye disorders) | 10 (11)
Conjunctival cyst (Eye disorders) | 2 (2)
Conjunctival dehiscence (Eye disorders) | 2 (2)
Conjunctival erosion (Eye disorders) | 2 (2)
Conjunctivitis - inflammatory (Eye disorders) | 4 (5)
Corneal abrasion (Eye disorders) | 1 (1)
Corneal dryness (Eye disorders) | 1 (1)
Corneal epithelial defect (Eye disorders) | 1 (1)
Corneal fold (Eye disorders) | 1 (1)
Corneal opacity (Eye disorders) | 1 (1)
Corneal Suture Broken (Eye disorders) | 2 (2)
Corneal vascularization (Eye disorders) | 2 (2)
Decrease in light perception (Eye disorders) | 1 (1)
Elective revision surgery (Eye disorders) | 7 (7) — Better placement of array on retina
Epiphora (Eye disorders) | 3 (3)
Epiretinal membrane (Eye disorders) | 11 (11)
Fibrosis around retinal tack (Eye disorders) | 2 (2)
Filamentary keratitis (Eye disorders) | 1 (1)
Foreign Body Sensation (Eye disorders) | 1 (2)
Headache (Eye disorders) | 3 (3) — Adjudicated as device related
High IOP (Eye disorders) | 2 (2)
Hyphema (Eye disorders) | 3 (3)
Hypotony (Eye disorders) | 7 (8)
Inflammation - ocular (Eye disorders) | 5 (5)
Irregular pupil (Eye disorders) | 1 (1)
Keratic Precipitates (Eye disorders) | 2 (3)
Nausea (General disorders) | 1 (1) — Adjudicated as device or procedure related
Nystagmus increase (Eye disorders) | 1 (1)
Ocular fibrin (Eye disorders) | 1 (1)
Pain - ocular (Eye disorders) | 9 (18)
Pre-retinal hemorrhage (Eye disorders) | 1 (1)
Proliferative Vitreoretinopathy (Eye disorders) | 1 (1)
Ptosis (Eye disorders) | 2 (2)
Retinal Break/Tear (Eye disorders) | 1 (1)
Retinal detachment - tractional (Eye disorders) | 1 (1)
Retinal folds (Eye disorders) | 1 (1)
Retinal Thickening - cystoid macular edema (CME) (Eye disorders) | 4 (4)
Retinal Thickening - without cystic changes (Eye disorders) | 4 (4)
Retinoschisis (Eye disorders) | 1 (2)
Revision Surgery - tack replacement (Eye disorders) | 1 (1)
Rubeosis (Eye disorders) | 1 (1)
Scleral graft displacement or reabsorption (Eye disorders) | 2 (2)
Scleritis (Eye disorders) | 1 (1)
Suture irritation (General disorders) | 6 (7) — Associated with surgical procedure
Uveitis (Eye disorders) | 5 (6)
Vertigo (General disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-01-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT00407602/Prot_SAP_ICF_000.pdf